CLINICAL TRIAL: NCT02287207
Title: Effects of Transcranial Direct Current Stimulation on Fine Motor Skills in Parkinson's Disease: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Alice Nieuwboer, Professor, KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: S57231
Record Dates: First submitted 2014-11-03; First posted 2014-11-10 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2015-11

CONDITIONS: Parkinson's Disease; Transcranial Direct Current Stimulation; Fine Motor Skills; Handwriting
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Anodal tDCS (Active Comparator): 20 minutes, 1.0 mA unilateral-anodal motor cortex (M1) tDCS stimulation
  Interventions: Device: transcranial direct current stimulation (tDCS)
- Sham tDCS (Sham Comparator): 20 minutes, sham tDCS stimulation
  Interventions: Device: transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: transcranial direct current stimulation (tDCS)

SUMMARY:
The purpose of this pilot study is to determine the effect of transcranial direct current stimulation (tDCS) on brain activity and fine motor skills in patients with Parkinson's disease compared to healthy controls.

DETAILED DESCRIPTION:
The pilot study will involve a double-blind, sham controlled cross-over design where participants will receive anodal and sham tDCS stimulation in a randomized order. Differences in brain activity and fine motor skill performance between groups and after tDCS stimulation will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with idiopathic PD, according to the UK Brain Bank criteria
* Hoehn and Yahr (H&Y) stage II in the 'on'-phase of the medication cycle
* Right dominant PD

Exclusion Criteria:

* Cognitive impairment (MMSE < 23)
* Visuo-spatial deficits (measured by the Rey-Osterrieth Complex Figure (ROCF) test)
* Left-handedness (evaluated by the Edinburgh Handedness scale)
* Depression
* Pregnancy
* Alcohol abuse
* Aneurysm clips
* Pacemaker
* Neurostimulator
* Implemented defibrillator
* Magnetically activated implant or device
* Implemented pump
* Spinal cord simulator
* Implemented hearing aid
* Artificial or prosthetic limb
* Metal parts in the body
* Any external or internal metal
* Artificial heart valve
* Other implants
* History of brain surgery
* Migraine
* Family history of Epilepsy
* Other contra-indications for tDCS and Transcranial Magnetic Stimulation (TMS)
* Other neurological, psychiatric or interfering upper limb problems

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change in writing amplitude | post-stimulation (immediately after) and retention (1 week)
  Centimeter (cm)
Change in writing velocity | post-stimulation (immediately after) and retention (1 week)
  Centimeter per second (cm/s)

SECONDARY OUTCOMES:
Change in speed on the Purdue Pegboard task | post-stimulation (immediately after) and retention (1 week)
  Number of pegs placed in 30 seconds
Change in cortical excitability | post-stimulation (immediately after) and retention (1 week)
  Motor Evoked Potentials (MEP) peak to peak amplitude and latency - Measured with single-pulse Transcranial Magnetic
Change in Short-Latency Intracortical Inhibition (SICI) | post-stimulation (immediately after) and retention (1 week)
  Measured with double-pulse Transcranial Magnetic Stimulation (TMS)
Change in cortical silent period (cSP) | post-stimulation (immediately after) and retention (1 week)
  Measured with single-pulse Transcranial Magnetic

CONTACTS AND LOCATIONS:
Locations (1):
- CatholicULeuven, Leuven, Belgium

REFERENCES:
- [Background] Broeder S, Nackaerts E, Nieuwboer A, Smits-Engelsman BC, Swinnen SP, Heremans E. The effects of dual tasking on handwriting in patients with Parkinson's disease. Neuroscience. 2014 Mar 28;263:193-202. doi: 10.1016/j.neuroscience.2014.01.019. Epub 2014 Jan 19. PMID 24447597
- [Background] Nackaerts E, Vervoort G, Heremans E, Smits-Engelsman BC, Swinnen SP, Nieuwboer A. Relearning of writing skills in Parkinson's disease: a literature review on influential factors and optimal strategies. Neurosci Biobehav Rev. 2013 Mar;37(3):349-57. doi: 10.1016/j.neubiorev.2013.01.015. Epub 2013 Jan 16. PMID 23333265
- [Background] Broeder S, Nackaerts E, Heremans E, Vervoort G, Meesen R, Verheyden G, Nieuwboer A. Transcranial direct current stimulation in Parkinson's disease: Neurophysiological mechanisms and behavioral effects. Neurosci Biobehav Rev. 2015 Oct;57:105-17. doi: 10.1016/j.neubiorev.2015.08.010. Epub 2015 Aug 20. PMID 26297812
- See also: Neuromotor Rehabilitation Research Group - KU Leuven, Belgium — http://gbiomed.kuleuven.be/english/research/50000743/nrrg1/nrrg.htm